Last updated: June 24, 2022

Mindfulness-based Queer Resilience (MBQR) to Promote Mental and Sexual Health among Sexual and Gender Minority Young Adults: Statistical Analysis Plan

A mixed-methods approach will be used to understand feasibility, acceptability, and longitudinal effects of this single-arm clinical trial. Descriptive statistics will be used to summarize feasibility and acceptability measures from the full sample. These measures include recruitment rates, retention/attrition rates, session attendance, Client Satisfaction Questionnaire, and session evaluation form.

In addition, qualitative data from exit interviews will be analyzed using template analysis, a thematic analysis methodology that applies data reduction techniques for rapid turnaround, often used in intervention development and refinement research.